CLINICAL TRIAL: NCT00715221
Title: Multi-Tracer Pet Quantitation of Insulin Action
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Padova (Other)
Responsible Party: Principal Investigator, Bret Goodpaster, Professor of Medicine, University of Pittsburgh
Other Study IDs: PRO 07080301
Record Dates: First submitted 2008-07-10; First posted 2008-07-15 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Diabetes
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Aliquotted blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Normal Weight
- 2: Obese without diabetes
- 3: Obese with diabetes

SUMMARY:
We are proposing a clinical investigation of the pathogenesis of insulin resistance (IR) in skeletal muscle and adipose tissue (AT), focusing specifically on the contributions of glucose delivery, transport and phosphorylation. The primary methodology will be dynamic PET imaging, using three tracers that respectively portray the kinetics of glucose delivery, bi-directional trans-membrane glucose transport and glucose phosphorylation. The three tracers are: 1) [15O]-H2O for quantifying tissue perfusion, this portrays the kinetics of glucose delivery from plasma to tissue; 2) [11C]-3-O-methyl glucose, a tracer constrained to bi-directional trans-membrane glucose transport; and 3) [18F]-fluoro-deoxy glucose, which like [11C]-3-OMG is transported, but adds the subsequent metabolic step, that of glucose phosphorylation.

We propose 2 specific aims to apply this methodology to investigate the pathogenesis of IR. The 1st aim is to quantitatively assess the kinetics of glucose delivery, transport and phosphorylation in skeletal muscle in type 2 DM and as compared to obese and lean non-diabetic men and women. We will appraise the contribution of each step to the to the pathogenesis of IR. We postulate more severe IR in oxidative muscle, with a dual impairment of glucose transport and phosphorylation. The 2nd aim is to implement the triple-tracer dynamic PET imaging protocol in adipose tissue (AT), examining normal insulin action in non-obese volunteers and testing whether differences in AT insulin action are present in obese insulin sensitive volunteers compared to obese IR participants and the relation of AT IR to that of muscle and liver.

DETAILED DESCRIPTION:
We propose a clinical investigation of the pathogenesis of insulin resistance (IR) in skeletal muscle and adipose tissue (AT) in obesity and diabetes mellitus, focusing on the separate and interactive roles of glucose delivery, bi-directional trans-membrane glucose transport and glucose phosphorylation. The primary methodology will be dynamic PET imaging, using three tracers that respectively portray the kinetics of glucose delivery, transport and phosphorylation. The three tracers are: 1) [15O]-H2O for quantifying tissue perfusion, this parameter together with glucose concentration portrays the kinetics of glucose delivery from plasma to tissue interstitial space; 2) [11C]-3-O-methyl glucose, a tracer constrained to bi-directional trans-membrane glucose transport; and 3) [18F]-fluoro-deoxy glucose, which like [11C]-3-OMG is transported, but adds the subsequent metabolic step, that of glucose phosphorylation.

In our recently completed studies, we implemented this triple-tracer dynamic PET imaging protocol to investigate insulin action in lean, healthy individuals 1-3. Rates of glucose uptake can be obtained by other methods (e.g. the glucose clamp, arterio-venous limb balance). What is uniquely valuable with dynamic PET imaging is acquisition of a temporal plot of tracer uptake, one that is obtained within an organ rather than derived from plasma determinations. These tissue-time activity curves provide information to assess the velocity of metabolic steps. By doing this for each of the three tracers, assessment can be made of which among glucose delivery, transport and phosphorylation is rate-controlling, or more properly, how rate control is distributed amongst these steps. The triple-tracer procedure has provided novel, quantitative insight on the action of insulin to change this distribution of control, a re-distribution triggered in healthy individuals by robust activation of glucose transport. Robust activation of glucose transport increases permeability of muscle to glucose sufficiently that delivery manifests greater rate limitation than during basal conditions. Also, we have coupled PET bio-imaging with MRI to study specific muscles 1, 3. This approach has yielded provocative and unanticipated new findings. Unlike in lean non-diabetics, in whom oxidative muscle is more insulin sensitive (as widely demonstrated in animal studies), in type 2 and in type 1 DM, oxidative muscle is more severely IR. We are encouraged that this bio-imaging methodology will enable new insight into the pathogenesis of IR in skeletal muscle and that the approach can be successfully adapted for in vivo investigation of adipose tissue metabolism.

The 1st specific aim is to quantitatively assess the contribution of glucose delivery, transport and phosphorylation to the pathogenesis of skeletal muscle IR in type 2 DM and obesity.

The 2nd specific aim is to implement triple-tracer dynamic PET imaging to study insulin action in gluteal-femoral adipose tissue (GF-AT) of non-obese and obese women, investigating among the latter group mechanisms of IR of GF-AT, and the role that GF-AT IR may have in differentiating obese insulin-sensitive (OB-InS) from obese insulin-resistant (OB-IR) women.

Experiment Synopsis: During the past year, in pilot studies, we initiated PET imaging procedures for AT, using [18F]-FDG. We now propose full development of the triple tracer methodology in GF-AT. Non-obese and obese women will be studied, the latter recruited to form groups of obese insulin-sensitive (OB-IS) and obese insulin-resistant (OB-IR). Triple-tracer PET imaging will be done during basal and insulin stimulated conditions, using an infusion rate of 20 mU/min-m2. Complementary assessments will include: a) MRI and DXA to measure the quantity of fat-mass (FM), GF-AT, abdominal adipose depots (ABD-SAT and VAT); b) endogenous glucose production (EGP) assessed using a primed, constant infusion of [6,6] d2-glucose; c) an adipokine profile; and d) a needle biopsy of GF-AT for histological and other analyses.

ELIGIBILITY:
Inclusion Criteria:

Male and Female Normal Weight - non-diabetic (BMI 19-25) Overweight/Obese - non-diabetic (BMI 27-38) Type 2 DM (BMI 27-38)

Fasting lab glucose < 100 mg/dl (non-diabetic groups) HbA1c < 6.0 (non-diabetic group) HbA1c < 8.5 (diabetic group)

Ulnar artery patent bilaterally Negative urine pregnancy test Non-smoker Independent in self blood glucose monitoring (diabetic group)

Exclusion Criteria:

BP > 150 mmHg systolic or > 95 mmHg diastolic History of any heart disease, including MI, pacemaker History of PVD, (including diminishing pulses) liver disease, kidney disease, pulmonary disease, neuromuscular disease, neurological disease, thyroid disease or any drug or alcohol abuse.

Current malignancy or history of cancer within the past 5 years Proteinuria 1+ or greater Hematocrit < 34% sTSH >8 ALT > 60; AST > 60; Alk Phos > 150 Total cholesterol > 250 Triglycerides > 300

MEDICATIONS:

Chronic medications that can alter glucose homeostasis: oral glucocorticoids, nicotinic acid (Birth control medications are okay and will not exclude) Thiazolidinediones or insulin, previous difficulty with lidocaine (xylocaine) Gained or lost more than 3 kg during the past 3 months Involved in regular exercise > 1 day/week Surgical or vascular implants, any metal in body, claustrophic Currently pregnant OR currently lactating

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Normal volunteer sample
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Physiological measurement; Differences in tissue insulin-stimulated glucose uptake used by PET imaging among normal weight, obese and patients with type 2 diabetes | Rate of glucose disposal during steady-state insulin stimulated conditions (hyperinsulinemia obtained via insulin infusions)
  PET-derived measures of muscle glucose uptake across three study groups - normal weight, obese and patients with type 2 diabetes (cross-sectional)

CONTACTS AND LOCATIONS:
Overall Officials: Bret H Goodpaster, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Goodpaster BH, Bertoldo A, Ng JM, Azuma K, Pencek RR, Kelley C, Price JC, Cobelli C, Kelley DE. Interactions among glucose delivery, transport, and phosphorylation that underlie skeletal muscle insulin resistance in obesity and type 2 Diabetes: studies with dynamic PET imaging. Diabetes. 2014 Mar;63(3):1058-68. doi: 10.2337/db13-1249. Epub 2013 Nov 12. PMID 24222345